CLINICAL TRIAL: NCT01720420
Title: A Clinical Evaluation of NobelProceraTM Implant Bar Overdenture in the Mandible or Maxilla on 4 NobelReplaceTM CC Implants
Brief Title: A Clinical Evaluation of NobelProcera Implant Bar Overdenture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nobel Biocare (Industry)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-174
Record Dates: First submitted 2012-10-22; First posted 2012-11-02 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Edentulous
Keywords: edentulous; maxilla; mandible; dental implant; bar; overdenture; Oral Health Impact Profile (OHIP); survival rate; technical complications; marginal bone level; soft tissue
MeSH Terms: conditions — Mouth, Edentulous | interventions — Denture, Overlay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mandible (Experimental): NobelReplace CC NobelProcera Implant Bar Titanium Overdenture (lab-made)
  Interventions: Device: NobelReplace CC, NobelProcera Implant Bar
- Maxilla (Experimental): NobelReplace CC NobelProcera Implant Bar Titanium Overdenture (lab-made)
  Interventions: Device: NobelReplace CC, NobelProcera Implant Bar

INTERVENTIONS:
Device: NobelReplace CC, NobelProcera Implant Bar — Implants titanium with conical connection, individualized titanium bar
  Other Names: NobelReplace CC implants; NobelProcera Implant Bar Titanium; Overdenture (lab-made)

SUMMARY:
AN OPEN 5-YEAR PROSPECTIVE, CLINICAL MULTI-CENTER STUDY on NobelProcera Implant Bar Titanium with Locator attachment and related Overdenture on 4 NobelReplace implants with conical connection (CC) in the mandible/maxilla.

DETAILED DESCRIPTION:
Study centers: 8 centers in 4 countries

Objectives of the study:

Primary Objective:

To evaluate and compare the clinical marginal bone level change (MBL) around the NobelReplaceTM CC implants supporting NobelProceraTM Implant Bar Overdenture (fixed-removable) in the mandible with the clinical marginal bone level change (MBL) of the NobelReplaceTM CC implants supporting NobelProceraTM Implant Bar Overdenture (fixed-removable) in the maxilla for a period of 5 years.

Secondary Objectives:

1. To evaluate and compare the cumulative survival rate (CSR) of the NobelReplaceTM CC implants supporting NobelProceraTM Implant Bar Overdenture (fixed-removable) in the mandible with the cumulative survival rate (CSR) of the NobelReplaceTM CC implants supporting NobelProceraTM Implant Bar Overdenture (fixed-removable) in the maxilla for a period of 5 years.
2. To evaluate and compare the cumulative survival rate (CSR) of NobelProceraTM Implant Bar Overdenture (fixed-removable) on four (4) NobelReplace CC implants in the mandible with the cumulative survival rate (CSR) of NobelProceraTM Implant Bar Overdenture (fixed-removable) on four (4) NobelReplace CC implants in the maxilla after 5 years.
3. To evaluate the clinical behaviour (soft tissue behavior, clinical function, patient satisfaction, Quality of Life and prosthetic maintenance needs such as wear, chipping of denture teeth, need for exchange of attachment components) of NobelProceraTM Implant Bar Overdenture (fixed-removable) in the mandible and maxilla over 5 years of clinical function.

Study design 5-year, open, prospective, clinical multi-center study.

Number of subjects 76 (in total), 7-9 per center

Patient population Adult female or male, at least 18 (or age of consent) and not older than 70 years, suitable for treatment with implant supported bar overdentures in the edentulous mandible or maxilla.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is at least 18 years of age (or age of consent) and has passed secession of growth
2. The subject is not older than 70 years
3. Obtained informed consent from the subject
4. Edentulous mandible or maxilla providing sufficient bone whereas removable NobelProceraTM Implant Bar Overdenture on four (4) implants is regarded as an appropriate treatment solution
5. The subject has an osseous architecture enough to receive four implants and a sufficient amount of bone for placing in healed or extraction sites implants with a length of at least 10mm
6. The implant site is free from infection and extraction remnants
7. Implants will be placed in healed or extractions sites, defined as a site with 8 weeks of healing following tooth extraction, respectively 6 months after major bone augmentation or soft tissue grafting
8. Good gingival / periodontal / periapical status of opposing teeth/implants
9. The subject fulfills the prerequisite that a harmonic, stable occlusal relationship can be achieved with opposing natural teeth resp. fixed or removable opposing dentition (tooth or implant based
10. The subjects as well as the implant site(s) fulfill the criteria for early loading (6 weeks until 3 months after implant placement)
11. The subject is in such a physical and mental condition that a 5-year follow-up period can be carried out without foreseeable problems
12. The subject is available for the 5-year term of the investigation
13. The subject is compliant with good oral hygiene

Exclusion Criteria:

1. The subject is not able to give her/his informed consent of participating
2. Health conditions, which do not permit the surgical (including anesthesia) or restorative procedure
3. Reason to believe that the treatment might have a negative effect on the subject's overall situation (psychiatric problems), as noted in subject records or in subject history
4. Any disorders in the planned implant area such as previous tumors, chronic bone disease or previous irradiation in the head/neck area
5. Alcohol or drug abuse as noted in subject records or in subject history
6. Smoking of >10 cigarettes/day
7. Uncontrolled diabetes, i.e. a subject with diagnosed diabetes that has a history of neglecting doctor's recommendations regarding treatment, food and alcohol intake
8. Pathologic occlusion, e.g. severe bruxism or other destructive habits
9. Lack of opposing dentition or unstable occlusion
10. Ongoing infections, endodontic or periodontal problems in opposing teeth or implants
11. Subject shows an unacceptable oral hygiene
12. Subject has allergic or adverse reactions to the restorative material.
13. Bone augmentation of more than 3mm vertical height performed less than 3 months prior to planned implant placement.
14. Long-term bis-phosphonate therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
MBL,marginal bone level change | 6 month, 1, 2, 3, 5 year
  To evaluate and compare the clinical marginal bone level change (change MBL)in relation to defined implant reference point and different time points in the maxilla and mandible(between baseline at implant insertion and follow-up time points at 1 month, 6 month, 1 year, 2 year, 3 year and 5 year after implant insertion) of observation.

SECONDARY OUTCOMES:
CSR implants | 6 month, 1, 2, 3, 5 year
  CSR in % of placed implants
CSR prosthetics | 6 month, 1, 2, 3, 5 year
  survival in % of placed final restorations
Gingival Status | 6 month, 1, 2, 3, 5 year
  Gingival status(Silness and Loe 1963):0 = Normal gingiva surrounding crown/control tooth,1 = Mild inflammation,2 = Moderate inflammation.3 = Severe inflammation.
Status of mucosa | 6 month, 1, 2, 3, 5 year,
  0 = No keratinized mucosa.1 = Mucosa partially keratinized.2 = entire mucosa keratinized.
Bleeding tendency | 6 month, 1, 2, 3, 5 year
  (modified Sulcus Bleeding Index_mBI)(Mombelli):0 = No bleeding when a periodontal probe is passed along gingival margin adjacent to the implant.1 = Isolated bleeding spots visible. 2 = Blood forms a confluent red line on the margin 3 = Heavy or profuse bleeding.
plaque accumulation | 6 month, 1, 2, 3, 5 year
  modified Plaque Index (mPlI) (Mombelli):0 = No detectible plaque. 1 = Plaque only recognized by running a probe across the marginal surface of the implant. 2 = Plaque can be seen by the naked eye.3 = Abundance of soft matter
Pocket depths | 6 month, 1, 2, 3, 5 year
  Pocket depths measured around implants in millimeter (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Heydecke, Prof, Principal Investigator — Poliklinik für Zahnärztliche Prothetik, University Hamburg; Alessandro Pozzi, Prof, Principal Investigator — University of Rome, Italy; Eugenio Romeo, Prof, Principal Investigator — University of Milan, Italy; Marco Ferrari, Prof, Principal Investigator — University of Siena, Italy; Edoardo Stellini, Prof, Principal Investigator — University of Padova, Italy; Nikolaus and Alexandra Behneke, Prof., Dr., Principal Investigator — University of Mainz, Germany; Silvio Meloni, Dr., Principal Investigator — Università degli Studi di Sassari
Locations (7):
- Germany (2):
  - Guido Heydecke, Hamburg
  - Nikolaus and Alexandra Behneke, Mainz
- Italy (5):
  - Eugenio Romeo, Milan
  - Edoardo Stellini, Padua
  - Alessandro Pozzi, Rome
  - Università degli Studi di Sassari, Sassari
  - Marco Ferrari, Siena